CLINICAL TRIAL: NCT03818035
Title: A Phase 3b, Randomized, Double-blind, Parallel Group, Multicenter Study to Evaluate Further Therapeutic Strategies With Guselkumab in Patients With Moderate-to-Severe Plaque-Type Psoriasis
Brief Title: A Study to Evaluate Further Therapeutic Strategies With Guselkumab in Participants With Moderate-to-Severe Plaque-Type Psoriasis
Acronym: GUIDE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen-Cilag International NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR108514; 2018-001238-16 (EudraCT Number); CNTO1959PSO3012 (Other: Janssen-Cilag International NV); 2023-508424-34-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2019-01-11; First posted 2019-01-28 (Actual); Results first posted 2023-05-10 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — guselkumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Part 1: Guselkumab (Experimental): Participants in group 1 (Part 1) will receive 100 milligram (mg) guselkumab subcutaneously (SC) at Weeks 0, 4, 12 and 20.
  Interventions: Drug: Guselkumab
- Part 2: Guselkumab q8w and Guselkumab q16w (Experimental): Eligible participants from Part 1 will continue to participate in Part 2. Participants (super responder [SRe]) with a Psoriasis Area and Severity Index (PASI) score = 0 at weeks 20 and 28 will be randomized to guselkumab 100 mg every 8 weeks (q8w) (group 2a) or guselkumab 100 mg q16w (group 2b), at weeks 28 to 60. Group 2b will receive placebo injection at weeks 28, 44 and 60 to keep the comparison double blind. Participants losing control of disease (PASI score >5) during study Part 2 (until week 60), will enter the re-treatment arm (group 2d) and receive guselkumab 100mg q8w (at re-treatment week 0), followed by administration at re-treatment-weeks 8 and 16.
  Interventions: Drug: Guselkumab
- Part 2: Guselkumab q8w (Experimental): Participants (Non SRe) in group 2c with a PASI score greater than (>) 0 at week 20 and/or 28 will continue to receive guselkumab 100 mg q8w until week 60.
  Interventions: Drug: Guselkumab; Drug: Placebo Injection
- Part 3: Guselkumab Withdrawal (Experimental): Participants from groups 2a and 2b with a PASI score <3 at week 68 will be included in Part 3 (group 3a and 3b) and be withdrawn from guselkumab. Study visits will be conducted every 12 weeks until week 220 (follow-up). Participants with fluctuating disease (PASI score greater than or equal to [>=] 3) at week 68 or PASI >5 (participants losing control of disease) at any visit during part 3 after week 68 will get an opportunity to enter the re-treatment-arm (group 3c) in which participants will receive three guselkumab injections of 100 mg q8w.
  Interventions: Drug: Guselkumab

INTERVENTIONS:
Drug: Guselkumab — Participants will receive 100 mg guselkumab subcutaneously at Weeks 0, 4, 12 and 20 (group 1), at weeks 28, 36, 44, 52, 60 (group 2a and 2c), and at weeks 36 and 52 (group 2b). Group 2d and 3c are the re-treatment groups and will receive three injections after loss of disease control.
  Other Names: TREMFYA
Drug: Placebo Injection — Participants of group 2b will receive matching placebo injection subcutaneously at weeks 28, 44 and 60.
  Arms: Part 2: Guselkumab q8w

SUMMARY:
The purpose of this study is to demonstrate that Super-Responders (SRe; defined as psoriasis participants who receive on-label guselkumab treatment until week 20 and respond with a Psoriasis Area and Severity Index score (PASI) = 0 at weeks 20 and 28) maintain control of disease until week 68 with prolonged treatment intervals of 16 weeks (guselkumab 100 mg every 16 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Has a disease duration of plaque psoriasis of either less than or equal to (<=2) years or (greater than (>2) years calculated from date at which first symptoms [plaque] were reported by subject to date of screening visit at screening; approximately 40 percentage (%) of participants must have a disease duration <=2 years
* Has moderate-to-severe plaque-psoriasis defined by a Psoriasis Area and Severity Index (PASI) score >10 or affected body surface area (BSA) >10%) and additionally a Dermatology Life Quality Index (DLQI) score >10 at baseline (week 0)
* Have no signs or symptoms suggestive of active tuberculosis (TB) upon medical history and/or physical examination
* Agrees not to receive a live virus or live bacterial vaccination during the study, or within 3 months after the last administration of study drug
* Agrees not to receive a Bacille Calmette-Guerin (BCG) vaccination during the study, or within 12 months after the last administration of study drug

Exclusion Criteria:

* Has previously received any therapeutic agent directly targeted to interleukin (IL) -23 (including but not limited to guselkumab, tildrakizumab [MK3222], risankizumab [BI-655066])
* Has received any systemic immunosuppressant (for example, methotrexate, azathioprine, cyclosporine, 6-thioguanine, mercaptopurine, mycophenolate mofetil, tacrolimus, fumaric acid esters), or anakinra within 4 weeks of the first administration of study drug.
* Tests positive for hepatitis B virus (HBV) infection or who are seropositive for antibodies to hepatitis C virus (HCV), unless they have 2 negative HCV RNA test results 6 months apart after completing antiviral treatment and prior to baseline and have a third negative HCV RNA test result at baseline
* Has received natalizumab, belimumab, or agents that modulate B cells or T cells (e.g., rituximab, alemtuzumab, abatacept, or visilizumab) within 12 months of the first administration of study drug
* Has received any anti - tumor necrosis factor (TNF)-α biologic therapy within 3 months before the first administration of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 880 (Actual)
Dates: Start 2019-02-08 (Actual); Primary Completion 2022-03-07 (Actual); Study Completion 2025-01-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag International NV Clinical Trial, Study Director — Janssen-Cilag International NV
Locations (89):
- France (11):
  - Hopital Prive d'Antony, Antony
  - Centre Hospitalier d'Auxerre, Auxerre
  - Polyclinique Reims Bezanne - De Courlancy, Bezanne
  - Centre Hospitalier Le Mans, Le Mans
  - Hôpital Edouard Herriot, Lyon
  - Le Bateau Blanc, Martigues
  - CHU Nantes, Nantes
  - CHU de Nice Hopital de l Archet, Nice
  - CHU Rouen, Rouen
  - HIA se Sainte-Anne - Toulon, Toulon
  - CHU Toulouse, Toulouse
- Germany (78):
  - Universitätsklinikum Aachen, Aachen
  - DermaManagement Augsburg GmbH, Augsburg
  - Klinikum Augsburg, Augsburg
  - Fachklinik Bad Bentheim, Bad Bentheim
  - Hautmedizin Bad Soden, Bad Soden am Taunus
  - Charite CCM, Dermatologie, Berlin
  - Vivantes Klinikum Im Friedrichshain, Berlin
  - Rothhaar Studien GmbH, Berlin
  - ISA - Interdisciplinary Study Association GmbH, Berlin
  - Hautarztpraxis, Berlin
  - Hautarztpraxis Dr.Wildfeuer, Berlin
  - Praxis 'Haut Pur', Berlin
  - Klinikum Bielefeld Rosenhoehe, Bielefeld
  - Katholisches Klinikum Bochum gGmbH, Bochum
  - Niesmann & Othlinghaus GbR, Bochum
  - MVZ Dermatologisches Zentrum Bonn GmbH, Bonn
  - Universitatsklinikum Bonn, Bonn
  - Hautarztpraxis, Borna
  - Hautarztpraxis, Bramsche
  - Derma Nord, Bremen
  - Universitaetsklinikum Koeln, Cologne
  - Klinikum Darmstadt GmbH - Hautklinik, Darmstadt
  - Rosenpark Research GmbH, Darmstadt
  - Klinische Forschung Dresden GmbH, Dresden
  - Praxis für Dermatologie und Venerologie, Dresden
  - University Hospital Dresden, Dresden
  - Pro Derma, Dülmen
  - Privatpraxis Dr. Hilton & Partner, Düsseldorf
  - Universitatsklinikum Dusseldorf, Düsseldorf
  - Universitaetsklinik Erlangen, Erlangen
  - Universitaetsklinikum Essen, Essen
  - Universitatsklinikum Frankfurt, Frankfurt am Main
  - Universitatsklinikum Freiburg, Freiburg im Breisgau
  - Derma-Study-Center Friedrichshafen GmbH, Friedrichshafen
  - SRH Waldklinikum Gera GmbH, Gera
  - Hautarztpraxis Brau/Groß, Giessen
  - Universitatsmedizin Gottingen, Göttingen
  - Universitaetsklinik Hamburg-Eppendorf, Hamburg
  - Klinische Forschung Hamburg, Hamburg
  - Dermatologikum Hamburg Gmbh, Hamburg
  - SCIderm GmbH, Hamburg
  - MensingDerma research GmbH, Hamburg
  - Die Hautklinik Hanau, Hanau
  - Haut- und Laserzentrum Heidelberg, Heidelberg
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Hautarztpraxis Offers/Adamini, Ibbenbueren
  - Universitatsklinikum Jena, Jena
  - Universitatsklinikum Schleswig Holstein Kiel, Kiel
  - MVZ DermaKiel GmbH, Kiel
  - Praxis Dr. med. Beate Schwarz - Germany, Langenau
  - Universitatsklinikum Leipzig AOR, Leipzig
  - Hautarztpraxis, Lingen
  - Otto Von Guericke Universität Magdeburg, Magdeburg
  - Gemeinschaftspraxis Scholz/Sebastian/Schilling, Mahlow
  - Hautarztzentrum am MDZ, Mainz
  - Universitaetsmedizin Mainz, Mainz
  - Universitaetsklinikum Mannheim, Mannheim
  - Hautarztpraxis, Memmingen
  - Zentderma BAG Dres. Ostendorf - Bohm - Jo GbR, Mönchengladbach
  - Technische Universitaet Muenchen, München
  - Universitaetsklinikum Muenster, Münster
  - Klinikum Oldenburg, Oldenburg
  - Klinische Forschung Osnabrück, Osnabrück
  - Hautarztpraxis, Potsdam
  - Harzklinikum Dorothea Christiane Erxleben GmbH - Germnay, Quedlinburg
  - Universitaetsklinikum Regensburg, Regensburg
  - Hautarztpraxis Mortazawi, Remscheid
  - Klinische Forschung Schwerin GmbH, Schwerin
  - Company for Medical Study & Service Selters, Selters
  - Hautarztpraxis Dr. Leitz & Kollegen, Stuttgart
  - Hautarztpraxis am Loewenmarkt, Stuttgart
  - Universitatsklinikum Tubingen, Tübingen
  - Universitatsklinikum Ulm, Ulm
  - Hautarztpraxis Kock, Vechta
  - Centrovital, Witten
  - HELIOS Klinikum Wuppertal GmbH, Wuppertal
  - CentroDerm GmbH, Wuppertal
  - Universitatsklinikum Wurzburg, Würzburg

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Eyerich K, Asadullah K, Pinter A, Weisenseel P, Reich K, Paul C, Sabat R, Wolk K, Eyerich S, Lauffer F, Angsana J, Taut FJH, Kohler K, Chen Y, Sendecki J, Leung MWL, Wegner S, Personke Y, Gomez M, Kruger N, Tabori S, Schakel K. Noninferiority of 16-Week vs 8-Week Guselkumab Dosing in Super Responders for Maintaining Control of Psoriasis: The GUIDE Randomized Clinical Trial. JAMA Dermatol. 2024 Sep 1;160(9):953-963. doi: 10.1001/jamadermatol.2024.2463. PMID 39083288
- [Derived] Eyerich K, Weisenseel P, Pinter A, Schakel K, Asadullah K, Wegner S, Munoz-Elias EJ, Bartz H, Taut FJH, Reich K. IL-23 blockade with guselkumab potentially modifies psoriasis pathogenesis: rationale and study protocol of a phase 3b, randomised, double-blind, multicentre study in participants with moderate-to-severe plaque-type psoriasis (GUIDE). BMJ Open. 2021 Sep 13;11(9):e049822. doi: 10.1136/bmjopen-2021-049822. PMID 34518264

RESULTS

PARTICIPANT FLOW:
Groups:
- Part 1 Group 1: Guselkumab 100mg: Participants with moderate to severe plaque-type psoriasis received guselkumab 100 milligrams (mg) by subcutaneous (SC) injection at Weeks 0, 4, 12, and 20 in Part 1. Participants were followed from Week 0 through Week 28 or early termination prior to Week 28.
- Part 2 Group 2a: Guselkumab 100 mg Q8W: Super responders (SRe) (Psoriasis Area and Severity Index [PASI] score = 0 at Week 20 and Week 28) who completed study Part 1, were randomized to receive guselkumab 100 mg by SC injection every 8 weeks (Q8W) starting at Week 28 until Week 60. Participants were followed from Week 28 until Week 68 or early termination prior to Week 68.
- Part 2 Group 2b: Guselkumab 100 mg Q16W: Super responders (PASI score = 0 at Week 20 and Week 28) who completed study Part 1, were randomized to receive guselkumab 100 mg by SC injection every 16 weeks (Q16W) at Weeks 36 and 52. To maintain the study blind, participants were administered placebo by SC injection at Weeks 28, 44 and 60. Participants were followed from Week 28 until Week 68 or early termination prior to Week 68.
- Part 2 Group 2c: Guselkumab 100 mg Q8W: Non-super responders (PASI score greater than [>] 0 at Week 20 and/or Week 28) who completed study Part 1 continued to receive guselkumab 100 mg by SC injection Q8W starting at Week 28 until Week 60. Participants were followed from Week 28 until Week 68 or early termination prior to Week 68.
- Part 2 Group 2d: Re-Treatment Guselkumab 100mg: Participants from Groups 2a and 2b who lost control of disease (PASI >=5) until Week 60 or were not eligible to enter withdrawal (PASI >=3) at Week 68 were re-treated as Group 2d, receiving guselkumab 100 mg by SC injection at re-treatment Weeks 0, 8, and 16 from entering Group 2d.
- Part 3 Group 3a: Withdrawal (Q8W): Super responders from Group 2a with PASI score <= 3 were withdrawn from guselkumab 100 mg at Week 68. Participants were followed until Week 220.
- Part 3 Group 3b: Withdrawal (Q16W): Super responders from Group 2b with PASI score <= 3 were withdrawn from guselkumab 100 mg at Week 68. Participants were followed until Week 220.
- Part 3 Group 3c: Re-Treatment Guselkumab 100mg: Super responders with loss of disease control at or any visit after Week 68 who entered the re-treatment (R) arm and received guselkumab 100 mg by SC injection at re-treatment Weeks 0, 8 and 16 calculated from the date of loss of disease control. Participants were followed from re-treatment Week 0 until re-treatment Week 28 calculated from start of re-treatment due to loss disease control.
Period: Part 1: Open-label (Week 0 to Week 8)
Arm/Group | Part 1 Group 1: Guselkumab 100mg | Part 2 Group 2a: Guselkumab 100 mg Q8W | Part 2 Group 2b: Guselkumab 100 mg Q16W | Part 2 Group 2c: Guselkumab 100 mg Q8W | Part 2 Group 2d: Re-Treatment Guselkumab 100mg | Part 3 Group 3a: Withdrawal (Q8W) | Part 3 Group 3b: Withdrawal (Q16W) | Part 3 Group 3c: Re-Treatment Guselkumab 100mg
Started | 880 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 822 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 58 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 11 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event - Worsening of Psoriasis | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event - Other | 16 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Non-Compliance with Study Drug | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2: Double-blind (Week28 to Week68)
Arm/Group | Part 1 Group 1: Guselkumab 100mg | Part 2 Group 2a: Guselkumab 100 mg Q8W | Part 2 Group 2b: Guselkumab 100 mg Q16W | Part 2 Group 2c: Guselkumab 100 mg Q8W | Part 2 Group 2d: Re-Treatment Guselkumab 100mg | Part 3 Group 3a: Withdrawal (Q8W) | Part 3 Group 3b: Withdrawal (Q16W) | Part 3 Group 3c: Re-Treatment Guselkumab 100mg
Started | 0 | 148 (Only eligible participants from Part 1, were randomized into Part 2.) | 150 (Only eligible participants from Part 1, were randomized into Part 2.) | 525 (All participants not eligible for randomization from Part 1 continued in Group 2c.) | 0 | 0 | 0 | 0
Treated | 0 | 148 | 149 | 525 | 0 | 0 | 0 | 0
Completed | 0 | 137 | 142 | 496 | 0 | 0 | 0 | 0
Not Completed | 0 | 11 | 8 | 29 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 6 | 1 | 9 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 8 | 0 | 0 | 0 | 0
Not completed — Other Adverse Events | 0 | 3 | 4 | 6 | 0 | 0 | 0 | 0
Not completed — Adverse Event, serious fatal | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Participants Started Retreatment Phase Within Study Part 2 before Week 68 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Period: Part3: Withdrawal (Week 68 to Week 220)
Arm/Group | Part 1 Group 1: Guselkumab 100mg | Part 2 Group 2a: Guselkumab 100 mg Q8W | Part 2 Group 2b: Guselkumab 100 mg Q16W | Part 2 Group 2c: Guselkumab 100 mg Q8W | Part 2 Group 2d: Re-Treatment Guselkumab 100mg | Part 3 Group 3a: Withdrawal (Q8W) | Part 3 Group 3b: Withdrawal (Q16W) | Part 3 Group 3c: Re-Treatment Guselkumab 100mg
Started | 0 | 0 | 0 | 0 | 0 | 136 | 137 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 7 | 6 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 129 | 131 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 9 | 3 | 0
Not completed — Other Adverse Events | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Non-compliance with study drug | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Not completed — Not Signed ICF | 0 | 0 | 0 | 0 | 0 | 5 | 4 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Retreatment started | 0 | 0 | 0 | 0 | 0 | 112 | 115 | 0
Period: Re-treatment (Week R0 Through Week R28)
Arm/Group | Part 1 Group 1: Guselkumab 100mg | Part 2 Group 2a: Guselkumab 100 mg Q8W | Part 2 Group 2b: Guselkumab 100 mg Q16W | Part 2 Group 2c: Guselkumab 100 mg Q8W | Part 2 Group 2d: Re-Treatment Guselkumab 100mg | Part 3 Group 3a: Withdrawal (Q8W) | Part 3 Group 3b: Withdrawal (Q16W) | Part 3 Group 3c: Re-Treatment Guselkumab 100mg
Started | 0 | 0 | 0 | 0 | 9 | 0 | 0 | 227
Completed | 0 | 0 | 0 | 0 | 9 (SRe participants with loss of disease control from Groups 2a and 2b, entered retreatment group 2d. Includes participants who were re-treated at Week 68.) | 0 | 0 | 219 (Includes participants who were re-treated after Week 68.)
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Other Adverse Events | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Part 1 Group 1: Guselkumab 100 mg: Participants with moderate to severe plaque-type psoriasis received guselkumab 100 milligrams (mg) by subcutaneous (SC) injection at Weeks 0, 4, 12, and 20 in Part 1. Participants were followed from Week 0 through Week 28 or early termination prior to Week 28.
Arm/Group | Part 1 Group 1: Guselkumab 100 mg
Number analyzed (Participants) | 880
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 817
  >=65 years | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.5 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 260
  Male | 620
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 8
  Black | 1
  White | 859
  More than one race | 2
  Unknown or Not Reported | 3
  Other | 7
Region of Enrollment [Count of Participants; unit: Participants]
  FRANCE | 52
  GERMANY | 828

OUTCOME MEASURES:

1. Primary Outcome: Group 2a and Group 2b: Percentage of Participants Who Achieved an Absolute Psoriasis Area and Severity Index (PASI) Score Less Than (<) 3 at Week 68
Description: Percentage of participants who achieved an absolute PASI <3 at Week 68 were reported. The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed separately for the percentage of the body surface area involved, which translates to a numeric score that ranged from 0 (indicated no involvement) to 6 (90 percent [%]-100% involvement), and for erythema, induration and scaling, which are each rated on a scale of 0 to 4. The PASI produces a numeric score that could range from 0 (no psoriasis) to 72 (maximum psoriasis). Higher score indicated greater severity of psoriasis.
Time Frame: Week 68
Population: For part 2, ITT analysis set included all randomized participants at week 28 or treated with at least one dose of study agent within study part 2 (study group 2c).
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Part 2 Group 2a: Guselkumab 100 mg Q8W | Part 2 Group 2b: Guselkumab 100 mg Q16W
Number analyzed (Participants) | 148 | 149
Percentage of participants | 92.6 [88.0 to 95.8] | 91.9 [87.3 to 95.3]
Statistical Analysis 1: Comparison: Part 2 Group 2a: Guselkumab 100 mg Q8W vs Part 2 Group 2b: Guselkumab 100 mg Q16W; Test type: Non-Inferiority — One-sided two-group normal approximation Wald Z-test with Mantel-Haenszel stratum weights for 'disease duration' to test for non-inferiority of 100 mg q16w to 100 mg q8w with non-inferiority margin of 10%. Stratified analysis results were reported; p = 0.0013, Wald Z-test; Risk Difference (RD) = -0.6, 90% CI 2-sided [-5.7 to 4.5]

2. Secondary Outcome: Groups 1 and 2c: Time to Improvement From Baseline (Week 0) in PASI Score
Description: Time to improvement from baseline in PASI 75/90/100 response for participants with short disease duration (SDD) and longer disease duration (LDD) was reported. PASI was used for assessing and grading severity of psoriatic lesions and their response to therapy. In PASI, body was divided into 4 regions: head, trunk, upper extremities, and lower extremities. Each of these areas was assessed separately for percentage of area involved, which translates to numeric score that ranged from 0 (no involvement) to 6 (90-100% involvement), and for erythema, induration, and scaling, which were each rated on a scale of 0 to 4. PASI produced numeric score ranging from 0 (no psoriasis) to 72 (maximum psoriasis). Higher score indicated more severe disease. PASI responders were participants with >=75%, >=90%, 100% improvement in PASI respectively. For Part 2, data is reported only for those groups in which participants had PASI improvement post Week 28.
Time Frame: Group 1: Week 0 up to Week 28; Group 2c: Week 28 up to Week 68
Population: ITT analysis set for part 1 included all participants treated with at least one dose of study agent. For part 2, ITT analysis set included all randomized participants at week 28 or treated with at least one dose of study agent within study part 2 (study group 2c).
Measure: Median (Inter-Quartile Range); unit: Days
Groups:
- Part 1 Group 1: Participants With Disease Duration <= 2 Years: All participants enrolled with psoriasis of <=2 years disease duration (Short Disease Duration, SDD) received guselkumab 100 mg by SC injection at Week 0, Week 4, Week 12, and Week 20. Participants were followed from Week 0 until Week 28 or until early termination prior to Week 28.
- Part 1 Group 1: Participants With Disease Duration > 2 Years: All participants enrolled with psoriasis of >2 years disease duration (Longer Disease Duration, LDD) received guselkumab 100 mg by SC injection at Week 0, Week 4, Week 12, and Week 20. Participants were followed from Week 0 until Week 28 or until early termination prior to Week 28.
- Part 2 Group 2c: Participants With Disease Duration <= 2 Years: Non Super responders (PASI score > 0 at Week 20 and/or Week 28) with psoriasis of <=2 years disease duration (SDD) who completed study part 1, received guselkumab 100 mg by SC injection every 8 weeks (Q8W) starting at Week 28 until Week 60. Participants were followed from Week 28 until Week 68 or early termination prior to Week 68.
- Part 2 Group 2c: Participants With Duration > 2 Years: Non Super responders (PASI score > 0 at Week 20 and/or Week 28) with psoriasis of >2 years disease duration (LDD) who completed study part 1, received guselkumab 100 mg by SC injection every 8 weeks (Q8W) starting at Week 28 until Week 60. Participants were followed from Week 28 until Week 68 or early termination prior to Week 68.
Arm/Group | Part 1 Group 1: Participants With Disease Duration <= 2 Years | Part 1 Group 1: Participants With Disease Duration > 2 Years | Part 2 Group 2c: Participants With Disease Duration <= 2 Years | Part 2 Group 2c: Participants With Duration > 2 Years
Number analyzed (Participants) | 357 | 523 | 178 | 347
Days
  PASI 75 | 84.0 [81.0 to 89.0] | 84.0 [81.0 to 90.0] | 84.0 [83.0 to 112.0] | 84.0 [83.0 to 105.0]
  PASI 90 | 89.0 [84.0 to 134.0] | 106.0 [84.0 to 140.0] | 112.0 [84.0 to 153.0] | 114.0 [84.0 to 196.0]
  PASI 100 | 141.0 [105.0 to 210.0] | 200.0 [113.0 to NA] — NA signifies that upper limit of Inter-quartile range was not estimable due to insufficient number of participants with events. | 308.0 [196.0 to 483.0] | 416.0 [198 to NA] — NA signifies that lower limit of Inter-quartile range was not estimable due to insufficient number of participants with events.

3. Secondary Outcome: Groups 1, 2a, 2b, 2c, 3a and 3b: Percentage of Participants With Short (<=2 Years) and Longer (>2 Years) Disease Duration Who Achieved an Absolute PASI Score of 0, <=1 and <3 at Weeks 20, 28, 68, 116, 164 and 220
Description: Percentage of participants with short (<=2 years) and longer (>2 years) disease duration who achieved an absolute PASI Score of 0, <=1 and less than (<) 3 was reported. PASI was a system used for assessing and grading severity of psoriatic lesions and their response to therapy. In PASI, body was divided into 4 regions: head, trunk, upper extremities, and lower extremities. Each of these areas was assessed separately for percentage of area involved, which translated to numeric score that ranged from 0 (indicated no involvement) to 6 (90%-100% involvement), and for erythema, induration, and scaling, which were each rated on a scale of 0 to 4. PASI produced a numeric score that could range from 0 (no psoriasis) to 72 (maximum psoriasis). Higher score indicated more severe disease.
Time Frame: Group 1: Weeks 20 and 28; Groups 2a, 2b, 2c: Week 68; Groups 3a and 3b: Weeks 116, 164 and 220
Population: ITT analysis set for part 1 included all participants treated with at least one dose of study agent. For part 2, ITT analysis set was used. Part 3, ITT set=all participants entering Part 3. N (overall number of participants analyzed)= number of participants evaluable for this outcome measure and 'n' (number analyzed)=number of participants analyzed at specified timepoints. n=0 signifies that timepoint was not applicable for that arm.
Measure: Number; unit: Percentage of participants
Groups:
- Part 2 Group 2a: Participants With Disease Duration <= 2 Years: Super responders (PASI score = 0 at Week 20 and Week 28) with psoriasis of <=2 years disease duration (SDD) who completed study Part 1, randomized to guselkumab 100 mg by SC injection every 8 weeks (Q8W) starting at Week 28 until Week 60. Participants were followed from Week 28 until Week 68 or early termination prior to Week 68.
- Part 2 Group 2a: Participants With Disease Duration > 2 Years: Super responders (PASI score = 0 at Week 20 and Week 28) with psoriasis of >2 years disease duration (LDD) who completed study Part 1, randomized to guselkumab 100 mg by SC injection every 8 weeks (Q8W) starting at Week 28 until Week 60. Participants were followed from Week 28 until Week 68 or early termination prior to Week 68.
- Part 2 Group 2b: Participants With Disease Duration <= 2 Years: Super responders (PASI score = 0 at Week 20 and Week 28) with psoriasis of <=2 years disease duration (SDD) who completed study part 1, randomized to guselkumab 100 mg by SC injection every 16 weeks received at Week 36 and Week 52, received placebo at Week 28, Week 44 and Week 60. Participants were followed from Week 28 until Week 68 or early termination prior to Week 68.
- Part 2 Group 2b: Participants With Disease Duration > 2 Years: Super responders (PASI score = 0 at Week 20 and Week 28) with psoriasis of >2 years disease duration (LDD) who completed study part 1, randomized to guselkumab 100 mg by SC injection every 16 weeks received at Week 36 and Week 52, received placebo at Week 28, Week 44 and Week 60. Participants were followed from Week 28 until Week 68 or early termination prior to Week 68.
- Part 2 Group 2c: Participants With Disease Duration > 2 Years: Non-Super responders (PASI score > 0 at Week 20 and/or Week 28) with psoriasis of >2 years disease duration (LDD) who completed study part 1, received guselkumab 100 mg by SC injection every 8 weeks starting at Week 28 until Week 60. Participants followed from Week 28 until Week 68 or early termination prior to Week 68.
- Part 3 Group 3a: Participants With Disease Duration <=2 Years: Super responders (PASI score < 3 at Week 68) with psoriasis of <=2 years disease duration (SDD) from Group 2a who were withdrawn from guselkumab 100 mg at Week 68. Participants were followed until Week 220.
- Part 3 Group 3a: Participants With Disease Duration> 2 Years: Super responders (PASI score < 3 at Week 68) with psoriasis of >2 years disease duration (LDD) from Group 2a who were withdrawn from guselkumab 100 mg at Week 68. Participants were followed until Week 220.
- Part 3 Group 3b: Participants With Disease Duration <= 2 Years: Super responders (PASI score < 3 at Week 68) with psoriasis of <=2 years disease duration (SDD) from Group 2b who were withdrawn from guselkumab 100 mg at Week 68. Participants were followed until Week 220.
- Part 3 Group 3b: Participants With Disease Duration > 2 Years: Super responders (PASI score < 3 at Week 68) with psoriasis of >2 years disease duration (LDD) from Group 2b who were withdrawn from guselkumab 100 mg at Week 68. Participants were followed until Week 220.
Arm/Group | Part 1 Group 1: Participants With Disease Duration <= 2 Years | Part 1 Group 1: Participants With Disease Duration > 2 Years | Part 2 Group 2a: Participants With Disease Duration <= 2 Years | Part 2 Group 2a: Participants With Disease Duration > 2 Years | Part 2 Group 2b: Participants With Disease Duration <= 2 Years | Part 2 Group 2b: Participants With Disease Duration > 2 Years | Part 2 Group 2c: Participants With Disease Duration <= 2 Years | Part 2 Group 2c: Participants With Disease Duration > 2 Years | Part 3 Group 3a: Participants With Disease Duration <=2 Years | Part 3 Group 3a: Participants With Disease Duration> 2 Years | Part 3 Group 3b: Participants With Disease Duration <= 2 Years | Part 3 Group 3b: Participants With Disease Duration > 2 Years
Number analyzed (Participants) | 357 | 523 | 75 | 73 | 76 | 73 | 178 | 347 | 67 | 69 | 71 | 66
Percentage of participants
  PASI = 0 (Week 20): number analyzed (Participants) | 357 | 523 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PASI = 0 (Week 20) | 49.3 | 32.7 |  |  |  |  |  |  |  |  |  |
  PASI <=1 (Week 20): number analyzed (Participants) | 357 | 523 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PASI <=1 (Week 20) | 67.8 | 54.3 |  |  |  |  |  |  |  |  |  |
  PASI <3 (Week 20): number analyzed (Participants) | 357 | 523 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PASI <3 (Week 20) | 85.2 | 82.4 |  |  |  |  |  |  |  |  |  |
  PASI = 0 ( Week 28): number analyzed (Participants) | 357 | 523 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PASI = 0 ( Week 28) | 51.8 | 39.4 |  |  |  |  |  |  |  |  |  |
  PASI <=1 (Week 28): number analyzed (Participants) | 357 | 523 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PASI <=1 (Week 28) | 70.3 | 59.5 |  |  |  |  |  |  |  |  |  |
  PASI <3 (Week 28): number analyzed (Participants) | 357 | 523 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PASI <3 (Week 28) | 86.8 | 83.9 |  |  |  |  |  |  |  |  |  |
  PASI = 0 (Week 68): number analyzed (Participants) | 0 | 0 | 75 | 73 | 76 | 73 | 178 | 347 | 0 | 0 | 0 | 0
  PASI = 0 (Week 68) |  |  | 81.3 | 80.8 | 73.7 | 64.4 | 39.9 | 37.2 |  |  |  |
  PASI <=1 (Week 68): number analyzed (Participants) | 0 | 0 | 75 | 73 | 76 | 73 | 178 | 347 | 0 | 0 | 0 | 0
  PASI <=1 (Week 68) |  |  | 86.7 | 93.2 | 81.6 | 76.7 | 73.6 | 55.9 |  |  |  |
  PASI <3 (Week 68): number analyzed (Participants) | 0 | 0 | 75 | 73 | 76 | 73 | 178 | 347 | 0 | 0 | 0 | 0
  PASI <3 (Week 68) |  |  | 90.7 | 94.5 | 93.4 | 90.4 | 88.8 | 79.8 |  |  |  |
  PASI = 0 (Week 116): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 67 | 69 | 71 | 66
  PASI = 0 (Week 116) |  |  |  |  |  |  |  |  | 14.9 | 4.3 | 12.7 | 1.5
  PASI <=1 (Week 116): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 67 | 69 | 71 | 66
  PASI <=1 (Week 116) |  |  |  |  |  |  |  |  | 25.4 | 5.8 | 18.3 | 3.0
  PASI <3 (Week 116): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 67 | 69 | 71 | 66
  PASI <3 (Week 116) |  |  |  |  |  |  |  |  | 34.3 | 11.6 | 26.8 | 10.6
  PASI = 0 (Week 164): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 67 | 69 | 71 | 66
  PASI = 0 (Week 164) |  |  |  |  |  |  |  |  | 10.4 | 1.4 | 5.6 | 0.0
  PASI <=1 (Week 164): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 67 | 69 | 71 | 66
  PASI <=1 (Week 164) |  |  |  |  |  |  |  |  | 13.4 | 1.4 | 7.0 | 0.0
  PASI <3 (Week 164): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 67 | 69 | 71 | 66
  PASI <3 (Week 164) |  |  |  |  |  |  |  |  | 14.9 | 2.9 | 12.7 | 3.0
  PASI = 0 (Week 220): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 67 | 69 | 71 | 66
  PASI = 0 (Week 220) |  |  |  |  |  |  |  |  | 9.0 | 0 | 5.6 | 0
  PASI <=1 (Week 220): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 67 | 69 | 71 | 66
  PASI <=1 (Week 220) |  |  |  |  |  |  |  |  | 9.0 | 0 | 5.6 | 0
  PASI <3 (Week 220): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 67 | 69 | 71 | 66
  PASI <3 (Week 220) |  |  |  |  |  |  |  |  | 10.4 | 0 | 7.0 | 1.5

4. Secondary Outcome: Group 3a and Group 3b: Percentage of Participants With Short (<=2 Years) and Longer (>2 Years) Disease Duration Who Retain Disease Control (Absolute PASI Score < 3)
Description: Percentage of participants who retain disease control (that is, absolute PASI score <3 from Week 68 through Week 220 for participants with short (<= 2 years) and longer (>2 years) disease duration was reported. Control of disease was defined as participants with a PASI score <3. PASI was a system used for assessing and grading severity of psoriatic lesions and their response to therapy. In PASI, body was divided into 4 regions: head, trunk, upper extremities, and lower extremities. Each of these areas was assessed separately for percentage of area involved, which translated to numeric score that ranged from 0 (indicated no involvement) to 6 (90%-100% involvement), and for erythema, induration, and scaling, which were each rated on a scale of 0 to 4. PASI produced a numeric score that could range from 0 (no psoriasis) to 72 (maximum psoriasis). Higher score indicated more severe disease
Time Frame: From Week 68 up to Week 220
Population: For part 3, ITT analysis set included all participants entering study part 3 (either group 3a or 3b).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part 3 Group 3a: Participants With Disease Duration <=2 Years | Part 3 Group 3a: Participants With Disease Duration> 2 Years | Part 3 Group 3b: Participants With Disease Duration <= 2 Years | Part 3 Group 3b: Participants With Disease Duration > 2 Years
Number analyzed (Participants) | 67 | 69 | 71 | 66
Percentage of participants | 7.5 [2.5 to 16.6] | 0.0 [0.0 to 5.2] | 2.8 [0.3 to 9.8] | 1.5 [0.0 to 8.2]

5. Secondary Outcome: Groups 1, 2a, 2b, 2c, 3a and 3b: Percentage of Participants Who Achieved a PASI 75/90/100 Response at Weeks 20, 28, 68, 116, 164, and 220
Description: Percentage of participants who achieved PASI 75/90/100 response were reported. PASI was a system used for assessing and grading severity of psoriatic lesions and their response to therapy. In PASI, body was divided into 4 regions: head, trunk, upper extremities, and lower extremities. Each of these areas was assessed separately for percentage of area involved, which translated to numeric score that ranged from 0 (indicated no involvement) to 6 (90%-100% involvement), and for erythema, induration, and scaling, which were each rated on a scale of 0 to 4. PASI produced a numeric score that could range from 0 (no psoriasis) to 72 (maximum psoriasis). Higher score indicated more severe disease. PASI 75 responders were defined as participants with >= 75% improvement in PASI from baseline. PASI 90 responders were defined as participants with >= 90% improvement in PASI from baseline. PASI 100 responders were defined as participants with 100% improvement in PASI from baseline.
Time Frame: Group 1: Weeks 20, 28; Groups 2a, 2b, 2c: Week 68; Groups 3a, 3b: Weeks 116, 164 and 220
Population: For part 1 and 2, ITT analysis set was used. For part 3, ITT analysis set included all participants entering study part 3. n=0 signifies that specific timepoint was not applicable for that arm. Here 'n' (number analyzed) signifies number of participants analyzed at specified timepoints
Measure: Number; unit: Percentage of participants
Arm/Group | Part 1 Group 1: Guselkumab 100mg | Part 2 Group 2a: Guselkumab 100 mg Q8W | Part 2 Group 2b: Guselkumab 100 mg Q16W | Part 2 Group 2c: Guselkumab 100 mg Q8W | Part 3 Group 3a: Withdrawal (Q8W) | Part 3 Group 3b: Withdrawal (Q16W)
Number analyzed (Participants) | 880 | 148 | 149 | 525 | 136 | 137
Percentage of participants
  PASI 75 (Week 20): number analyzed (Participants) | 880 | 0 | 0 | 0 | 0 | 0
  PASI 75 (Week 20) | 90.2 |  |  |  |  |
  PASI 75 (Week 28): number analyzed (Participants) | 880 | 0 | 0 | 0 | 0 | 0
  PASI 75 (Week 28) | 90.7 |  |  |  |  |
  PASI 90 (Week 20): number analyzed (Participants) | 880 | 0 | 0 | 0 | 0 | 0
  PASI 90 (Week 20) | 73.6 |  |  |  |  |
  PASI 90 (Week 28): number analyzed (Participants) | 880 | 0 | 0 | 0 | 0 | 0
  PASI 90 (Week 28) | 76.0 |  |  |  |  |
  PASI 100 (Week 20): number analyzed (Participants) | 880 | 0 | 0 | 0 | 0 | 0
  PASI 100 (Week 20) | 39.4 |  |  |  |  |
  PASI 100 (Week 28): number analyzed (Participants) | 880 | 0 | 0 | 0 | 0 | 0
  PASI 100 (Week 28) | 44.4 |  |  |  |  |
  PASI 75 (Week 68): number analyzed (Participants) | 0 | 148 | 149 | 525 | 0 | 0
  PASI 75 (Week 68) |  | 92.6 | 94.0 | 88.0 |  |
  PASI 90 (Week 68): number analyzed (Participants) | 0 | 148 | 149 | 525 | 0 | 0
  PASI 90 (Week 68) |  | 91.9 | 85.9 | 73.7 |  |
  PASI 100 (Week 68): number analyzed (Participants) | 0 | 148 | 149 | 525 | 0 | 0
  PASI 100 (Week 68) |  | 81.1 | 69.1 | 38.1 |  |
  PASI 75 (Week 116): number analyzed (Participants) | 0 | 0 | 0 | 0 | 136 | 137
  PASI 75 (Week 116) |  |  |  |  | 27.9 | 20.4
  PASI 75 (Week 164): number analyzed (Participants) | 0 | 0 | 0 | 0 | 136 | 137
  PASI 75 (Week 164) |  |  |  |  | 10.3 | 8.0
  PASI 75 (Week 220): number analyzed (Participants) | 0 | 0 | 0 | 0 | 136 | 137
  PASI 75 (Week 220) |  |  |  |  | 5.1 | 4.4
  PASI 90 (Week 116): number analyzed (Participants) | 0 | 0 | 0 | 0 | 136 | 137
  PASI 90 (Week 116) |  |  |  |  | 18.4 | 13.1
  PASI 90 (Week 164): number analyzed (Participants) | 0 | 0 | 0 | 0 | 136 | 137
  PASI 90 (Week 164) |  |  |  |  | 7.4 | 5.8
  PASI 90 (Week 220): number analyzed (Participants) | 0 | 0 | 0 | 0 | 136 | 137
  PASI 90 (Week 220) |  |  |  |  | 5.1 | 2.9
  PASI 100 (Week 116): number analyzed (Participants) | 0 | 0 | 0 | 0 | 136 | 137
  PASI 100 (Week 116) |  |  |  |  | 9.6 | 7.3
  PASI 100 (Week 164): number analyzed (Participants) | 0 | 0 | 0 | 0 | 136 | 137
  PASI 100 (Week 164) |  |  |  |  | 5.9 | 2.9
  PASI 100 (Week 220): number analyzed (Participants) | 0 | 0 | 0 | 0 | 136 | 137
  PASI 100 (Week 220) |  |  |  |  | 4.4 | 2.9

6. Secondary Outcome: Group 3a and Group 3b: Time to Loss of Disease Control (Absolute PASI Score >5) After Treatment Withdrawal
Description: Time to loss of disease control (absolute PASI score >5) after treatment withdrawal beyond Week 68 up to Week 220 were reported. PASI was a system used for assessing and grading severity of psoriatic lesions and their response to therapy. In PASI, body was divided into 4 regions: head, trunk, upper extremities, and lower extremities. Each of these areas was assessed separately for percentage of area involved, which translated to numeric score that ranged from 0 (indicated no involvement) to 6 (90%-100% involvement), and for erythema, induration, and scaling, which were each rated on a scale of 0 to 4. PASI produced a numeric score that could range from 0 (no psoriasis) to 72 (maximum psoriasis). Higher score indicated more severe disease.
Time Frame: From Week 68 up to Week 220
Population: For part 3, ITT analysis set included all participants entering study part 3 (either group 3a or 3b).
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Part 3 Group 3a: Withdrawal (Q8W) | Part 3 Group 3b: Withdrawal (Q16W)
Number analyzed (Participants) | 136 | 137
Days | 245 [203 to 286] | 189 [166 to 251]

7. Secondary Outcome: Group 1: Percentage of Participants With an Absolute PASI Score = 0 at Weeks 12, 16, 20 and 28
Description: Percentage of participants with an absolute PASI score = 0 at Weeks 12, 16, 20 and 28 were reported. PASI was a system used for assessing and grading severity of psoriatic lesions and their response to therapy. In PASI, body was divided into 4 regions: head, trunk, upper extremities, and lower extremities. Each of these areas was assessed separately for percentage of area involved, which translated to numeric score that ranged from 0 (indicated no involvement) to 6 (90%-100% involvement), and for erythema, induration, and scaling, which were each rated on a scale of 0 to 4. PASI produced a numeric score that could range from 0 (no psoriasis) to 72 (maximum psoriasis). Higher score indicated more severe disease.
Time Frame: Weeks 12, 16, 20 and 28
Population: ITT analysis set for part 1 included all participants treated with at least one dose of study agent.
Measure: Number; unit: Percentage of participants
Arm/Group | Part 1 Group 1: Guselkumab 100 mg
Number analyzed (Participants) | 880
Percentage of participants
  Week 12 | 17.8
  Week 16 | 29.0
  Week 20 | 39.4
  Week 28 | 44.4

8. Secondary Outcome: Groups 1, 2a, 2b, 2c, 3a, 3b and 3c: Change From Baseline (Week 0) in Dermatology Life Quality Index (DLQI) Score
Description: Change from baseline (Week 0) in DLQI score were reported. DLQI was a 10-item instrument questionnaire designed to assess the impact of the disease on a participant's quality of life. Each question was evaluated on a 4-point scale ranged from 0 (not at all) to 3 (very much); where higher scores indicated more impact on quality of life. Scores from all 10 questions added up to give DLQI total score ranged from 0 (not at all) to 30 (very much). Higher scores indicated more impact on quality of life of participants.
Time Frame: Group 1: Baseline (Week 0), Week 28; Group 2a, 2b, 2c: Baseline (Week 0), Week 68; Group 3a and Group 3b:Baseline (Week 0), Week 116, 164 and 220; Group 3c: Baseline (Re-Treatment [R] Week 0), Week R24
Population: For part 1 and 2 ITT analysis set was used. For part 3, ITT analysis set included all participants entering study part 3. Here 'n' (number analyzed) signifies number of participants analyzed at specified timepoints. n=0, signifies that specified timepoint was not applicable for that arm.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Part 1 Group 1: Guselkumab 100mg | Part 2 Group 2a: Guselkumab 100 mg Q8W | Part 2 Group 2b: Guselkumab 100 mg Q16W | Part 2 Group 2c: Guselkumab 100 mg Q8W | Part 3 Group 3a: Withdrawal (Q8W) | Part 3 Group 3b: Withdrawal (Q16W) | Part 3 Group 3c: Re-Treatment Guselkumab 100mg
Number analyzed (Participants) | 880 | 148 | 149 | 525 | 136 | 137 | 227
Score on scale
  Week 28: number analyzed (Participants) | 880 | 0 | 0 | 0 | 0 | 0 | 0
  Week 28 | -16.6 (6.2) |  |  |  |  |  |
  Week 68: number analyzed (Participants) | 0 | 148 | 149 | 525 | 0 | 0 | 0
  Week 68 |  | -18.8 (5.6) | -17.0 (5.5) | -17.1 (5.8) |  |  |
  Week 116: number analyzed (Participants) | 0 | 0 | 0 | 0 | 136 | 137 | 0
  Week 116 |  |  |  |  | -16.5 (6.3) | -15.5 (6.4) |
  Week 164: number analyzed (Participants) | 0 | 0 | 0 | 0 | 136 | 137 | 0
  Week 164 |  |  |  |  | -18.1 (6.7) | -17.4 (7.8) |
  Week 220: number analyzed (Participants) | 0 | 0 | 0 | 0 | 136 | 137 | 0
  Week 220 |  |  |  |  | -20.9 (6.0) | -16.3 (6.5) |
  Re-Treatment till R24 weeks: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 227
  Re-Treatment till R24 weeks |  |  |  |  |  |  | -10.1 (6.8)

9. Secondary Outcome: Groups 1, 2a, 2b, 2c, 3a, 3b and 3c: Percentage of Participants Who Achieved a DLQI Score 0/1 and <5
Description: Percentage of participants who achieved a DLQI score 0/1 and <5 was reported. DLQI was a 10-item instrument questionnaire designed to assess the impact of the disease on a participant's quality of life. Each question was evaluated on a 4-point scale ranged from 0 (not at all) to 3 (very much); where higher scores indicated more impact on quality of life. Scores from all 10 questions added up to give DLQI total score ranged from 0 (not at all) to 30 (very much). Higher scores indicated more impact on quality of life of participants.
Time Frame: Group 1: Week 28; Groups 2a, 2b, 2c: Week 68; Groups 3a and 3b: Week 116, 164 and 220; Group 3c: Week R24
Population: For part 1, 2 and 3 ITT analysis set was used. Here 'n' (number analyzed) signifies number of participants analyzed at specified timepoints. n=0 signifies that timepoint was not applicable for that arm.
Measure: Number; unit: Percentage of participants
Arm/Group | Part 1 Group 1: Guselkumab 100mg | Part 2 Group 2a: Guselkumab 100 mg Q8W | Part 2 Group 2b: Guselkumab 100 mg Q16W | Part 2 Group 2c: Guselkumab 100 mg Q8W | Part 3 Group 3a: Withdrawal (Q8W) | Part 3 Group 3b: Withdrawal (Q16W) | Part 3 Group 3a: Participants With Disease Duration <=2 Years | Part 3 Group 3a: Participants With Disease Duration> 2 Years | Part 3 Group 3b: Participants With Disease Duration <= 2 Years | Part 3 Group 3b: Participants With Disease Duration > 2 Years | Part 3 Group 3c: Re-Treatment Guselkumab 100mg
Number analyzed (Participants) | 880 | 148 | 149 | 525 | 136 | 137 | 67 | 69 | 71 | 66 | 227
Percentage of participants
  DLQI Score 0/1 (Week 28): number analyzed (Participants) | 880 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  DLQI Score 0/1 (Week 28) | 60.9 |  |  |  |  |  |  |  |  |  |
  DLQI Score<5 (Week 28): number analyzed (Participants) | 880 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  DLQI Score<5 (Week 28) | 78.4 |  |  |  |  |  |  |  |  |  |
  DLQI Score 0/1 (Week 68): number analyzed (Participants) | 0 | 148 | 149 | 525 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  DLQI Score 0/1 (Week 68) |  | 83.1 | 77.9 | 61.9 |  |  |  |  |  |  |
  DLQI Score<5 (Week 68): number analyzed (Participants) | 0 | 148 | 149 | 525 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  DLQI Score<5 (Week 68) |  | 89.2 | 85.2 | 78.9 |  |  |  |  |  |  |
  DLQI Score 0/1 (Week 116): number analyzed (Participants) | 0 | 0 | 0 | 0 | 136 | 137 | 0 | 0 | 0 | 0 | 0
  DLQI Score 0/1 (Week 116) |  |  |  |  | 15.4 | 10.9 |  |  |  |  |
  DLQI Score <5 (Week 116): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 67 | 69 | 71 | 66 | 0
  DLQI Score <5 (Week 116) |  |  |  |  |  |  | 34.3 | 15.9 | 26.8 | 7.6 |
  DLQI Score 0/1 (Week 164): number analyzed (Participants) | 0 | 0 | 0 | 0 | 136 | 137 | 0 | 0 | 0 | 0 | 0
  DLQI Score 0/1 (Week 164) |  |  |  |  | 8.1 | 5.8 |  |  |  |  |
  DLQI Score <5 (Week 164): number analyzed (Participants) | 0 | 0 | 0 | 0 | 136 | 137 | 0 | 0 | 0 | 0 | 0
  DLQI Score <5 (Week 164) |  |  |  |  | 8.1 | 8.0 |  |  |  |  |
  DLQI Score 0/1 (Week 220): number analyzed (Participants) | 0 | 0 | 0 | 0 | 136 | 137 | 0 | 0 | 0 | 0 | 0
  DLQI Score 0/1 (Week 220) |  |  |  |  | 4.4 | 2.9 |  |  |  |  |
  DLQI Score <5 (Week 220): number analyzed (Participants) | 0 | 0 | 0 | 0 | 136 | 137 | 0 | 0 | 0 | 0 | 0
  DLQI Score <5 (Week 220) |  |  |  |  | 5.1 | 4.4 |  |  |  |  |
  DLQI Score 0/1 RT24: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 227
  DLQI Score 0/1 RT24 |  |  |  |  |  |  |  |  |  |  | 73.1
  DLQI Score <5 RT24: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 227
  DLQI Score <5 RT24 |  |  |  |  |  |  |  |  |  |  | 87.7

10. Secondary Outcome: Groups 1, 2a, 2b, 2c, 3a, and 3b: Percent Change From Baseline (Week 0) in Psoriasis- Affected Body Surface Area (BSA)
Description: Percent change from baseline in the psoriasis affected BSA (%) was reported. The percentage of the psoriasis-affected BSA percentage is a system used for assessing the severity of psoriasis. The plaque coverage is estimated using the rule of palm (1 palm of the hand = 1% BSA)
Time Frame: Group 1: Baseline (Week 0), Week 12, 28; Group 2a, 2b, 2c: Baseline (Week 0), Week 52 and 68, Group 3a, 3b: Baseline (Week 0), Week 80, 104, 116, 140, 164, 188, 212 and 220
Population: For part 1, 2 and 3 ITT analysis set was used. Here, 'N' (overall number of participants analyzed) signifies number of participants evaluable for this outcome measure. Here 'n' (number analyzed) signifies number of participants analyzed at specified timepoints. n=0, signifies that specified timepoint was not applicable for that arm..
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Part 1 Group 1: Guselkumab 100mg | Part 2 Group 2a: Guselkumab 100 mg Q8W | Part 2 Group 2b: Guselkumab 100 mg Q16W | Part 2 Group 2c: Guselkumab 100 mg Q8W | Part 3 Group 3a: Withdrawal (Q8W) | Part 3 Group 3b: Withdrawal (Q16W)
Number analyzed (Participants) | 861 | 141 | 142 | 492 | 126 | 107
Percent Change
  At Week 12: number analyzed (Participants) | 839 | 0 | 0 | 0 | 0 | 0
  At Week 12 | -19.3 (14.2) |  |  |  |  |
  At Week 28: number analyzed (Participants) | 861 | 0 | 0 | 0 | 0 | 0
  At Week 28 | -23.8 (15.0) |  |  |  |  |
  At Week 52: number analyzed (Participants) | 0 | 141 | 142 | 492 | 0 | 0
  At Week 52 |  | -25.1 (15.1) | -24.3 (15.6) | -24.8 (14.6) |  |
  At Week 68: number analyzed (Participants) | 0 | 136 | 137 | 492 | 0 | 0
  At Week 68 |  | -24.8 (14.9) | -24.3 (15.8) | -25.0 (14.6) |  |
  At Week 80: number analyzed (Participants) | 0 | 0 | 0 | 0 | 126 | 107
  At Week 80 |  |  |  |  | -23.8 (14.1) | -23.6 (15.6)
  At Week 104: number analyzed (Participants) | 0 | 0 | 0 | 0 | 54 | 45
  At Week 104 |  |  |  |  | -20.6 (15.1) | -22.5 (16.8)
  At Week 116: number analyzed (Participants) | 0 | 0 | 0 | 0 | 42 | 31
  At Week 116 |  |  |  |  | -22.4 (16.8) | -19.8 (13.0)
  At Week 140: number analyzed (Participants) | 0 | 0 | 0 | 0 | 18 | 14
  At Week 140 |  |  |  |  | -16.7 (8.5) | -19.6 (11.2)
  At Week 164: number analyzed (Participants) | 0 | 0 | 0 | 0 | 14 | 12
  At Week 164 |  |  |  |  | -18.2 (8.7) | -20.6 (11.2)
  At Week 188: number analyzed (Participants) | 0 | 0 | 0 | 0 | 11 | 7
  At Week 188 |  |  |  |  | -18.1 (8.2) | -20.4 (13.0)
  At Week 212: number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 6
  At Week 212 |  |  |  |  | -18.3 (9.6) | -19.3 (13.9)
  At Week 220: number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 6
  At Week 220 |  |  |  |  | -18.3 (9.6) | 19.0 (13.6)

11. Secondary Outcome: Groups 1, 2a, 2b, 2c, 3a and 3b: Change From Baseline in Nail Assessment in Psoriasis and Psoriatic Arthritis- Clinical (NAPPA-CLIN) at Weeks 28, 68, 116, 164 and 220
Description: Change from baseline in NAPPA-CLIN at Weeks 28, 68, 116 164, and 220 was reported. NAPPA-CLIN is an instrument used by the physician to assess the least and the worst involved nail of both hands or both feet with scores ranging from 0 (no involvement) to 16 (worst involvement). A higher score indicated a worst involvement.
Time Frame: Group 1: Baseline (Week 0), Week 28; Group 2a, 2b, 2c: Baseline (Week 0), Week 68; Group 3a and Group 3b: Baseline (Week 0), Week 116, 164, and 220
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Part 1 Group 1: Guselkumab 100mg | Part 2 Group 2a: Guselkumab 100 mg Q8W | Part 2 Group 2b: Guselkumab 100 mg Q16W | Part 2 Group 2c: Guselkumab 100 mg Q8W | Part 3 Group 3a: Withdrawal (Q8W) | Part 3 Group 3b: Withdrawal (Q16W)
Number analyzed (Participants) | 406 | 59 | 60 | 276 | 10 | 11
Score on scale
  Hands (Week 28): number analyzed (Participants) | 406 | 0 | 0 | 0 | 0 | 0
  Hands (Week 28) | -3.4 (3.2) |  |  |  |  |
  Feet (Week 28): number analyzed (Participants) | 352 | 0 | 0 | 0 | 0 | 0
  Feet (Week 28) | -3.1 (3.5) |  |  |  |  |
  Hands (Week 68): number analyzed (Participants) | 0 | 59 | 60 | 276 | 0 | 0
  Hands (Week 68) |  | -4.0 (3.2) | -4.5 (3.5) | -4.0 (3.2) |  |
  Feet (Week 68): number analyzed (Participants) | 0 | 46 | 48 | 250 | 0 | 0
  Feet (Week 68) |  | -4.9 (3.5) | -4.6 (3.7) | -4.1 (3.6) |  |
  Hands (Week 116): number analyzed (Participants) | 0 | 0 | 0 | 0 | 10 | 11
  Hands (Week 116) |  |  |  |  | -2.2 (4.3) | -2.2 (3.2)
  Feet (Week 116): number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 10
  Feet (Week 116) |  |  |  |  | -3.4 (6.2) | -3.5 (3.9)
  Hands (Week 164): number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 4
  Hands (Week 164) |  |  |  |  | -4.5 (3.5) | -3.0 (2.4)
  Feet (Week 164): number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 5
  Feet (Week 164) |  |  |  |  | -8.0 (NA) — 'NA' signifies that SD could could not be calculated for a single participant. | -3.6 (3.1)
  Hands (Week 220): number analyzed (Participants) | 0 | 0 | 0 | 0 | 3 | 3
  Hands (Week 220) |  |  |  |  | -4.3 (2.5) | -3.7 (2.5)
  Feet (Week 220): number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 4
  Feet (Week 220) |  |  |  |  | -8.0 (NA) — 'NA' signifies that SD could could not be calculated for a single participant. | -4.0 (3.5)

12. Secondary Outcome: Groups 1, 2a, 2b, 2c, 3a and 3b: Change From Baseline (Week 0) in the Signs and Symptoms Aggregate Scores of the Psoriasis Symptoms and Signs Diary (PSSD) at Weeks 28, 68, 116, 164 and 220
Description: Change from baseline (Week 0) in the signs and symptoms aggregate scores of the PSSD at Weeks 28, 68, 116, 164 and 220 was reported. The PSSD was a questionnaire designed to measure the severity of psoriasis symptoms and signs for the assessment of treatment benefit. PSSD was a participant self-administered outcomes instrument that included 11 items covering symptoms (itch, pain, stinging, burning and skin tightness) and participant observable signs (skin dryness, cracking, scaling, shedding or flaking, redness and bleeding) using 0 to 10 numerical rating scales for severity. Two sub scores each ranging from 0 to 100 were derived: the psoriasis symptom score and the psoriasis sign score. A higher score indicated more severe disease. A change of >= 40 points in PSSD symptom score or sign score, and a >= 3-point change in individual PSSD item scale scores was defined as clinically meaningful change (response).
Time Frame: as for outcome 11
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Part 1 Group 1: Guselkumab 100mg | Part 2 Group 2a: Guselkumab 100 mg Q8W | Part 2 Group 2b: Guselkumab 100 mg Q16W | Part 2 Group 2c: Guselkumab 100 mg Q8W | Part 3 Group 3a: Withdrawal (Q8W) | Part 3 Group 3b: Withdrawal (Q16W)
Number analyzed (Participants) | 863 | 138 | 140 | 492 | 41 | 31
Score on scale
  At Week 28 (Symptom): number analyzed (Participants) | 863 | 0 | 0 | 0 | 0 | 0
  At Week 28 (Symptom) | -57.2 (25.4) |  |  |  |  |
  At Week 28 (Sign): number analyzed (Participants) | 863 | 0 | 0 | 0 | 0 | 0
  At Week 28 (Sign) | -62.1 (22.0) |  |  |  |  |
  At Week 68 (Symptom): number analyzed (Participants) | 0 | 138 | 140 | 492 | 0 | 0
  At Week 68 (Symptom) |  | -65.1 (21.2) | -58.7 (23.3) | -58.6 (25.1) |  |
  At Week 68 (Sign): number analyzed (Participants) | 0 | 138 | 140 | 492 | 0 | 0
  At Week 68 (Sign) |  | -71.7 (16.4) | -65.4 (19.6) | -63.0 (22.2) |  |
  At Week 116 (Symptom): number analyzed (Participants) | 0 | 0 | 0 | 0 | 41 | 31
  At Week 116 (Symptom) |  |  |  |  | -52.3 (25.7) | -50.0 (24.3)
  At Week 116 (Sign): number analyzed (Participants) | 0 | 0 | 0 | 0 | 41 | 31
  At Week 116 (Sign) |  |  |  |  | -56.1 (25.6) | -52.2 (24.3)
  At Week 164 (Symptom): number analyzed (Participants) | 0 | 0 | 0 | 0 | 14 | 12
  At Week 164 (Symptom) |  |  |  |  | -59.7 (20.5) | -54.0 (26.1)
  At Week 164 (Sign): number analyzed (Participants) | 0 | 0 | 0 | 0 | 14 | 12
  At Week 164 (Sign) |  |  |  |  | -62.1 (22.0) | -50.4 (26.5)
  At Week 220 (Symptom): number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 6
  At Week 220 (Symptom) |  |  |  |  | -56.0 (22.9) | -54.7 (23.1)
  At Week 220 (Sign): number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 6
  At Week 220 (Sign) |  |  |  |  | -63.3 (20.3) | -54.7 (28.5)

13. Secondary Outcome: Groups 2a, 2b and 2c: Percentage of Participants Who Achieved a PSSD Sign Score = 0 at Week 68 in Participants With a PSSD Sign Score >= 1 at Week 28
Description: Percentage of participants who achieved a PSSD sign score = 0 at Week 68 in participants with a PSSD sign score >= 1 at Week 28 was reported. The PSSD was a questionnaire designed to measure the severity of psoriasis symptoms and signs for the assessment of treatment benefit. PSSD was a participant self-administered outcomes instrument that included 11 items covering symptoms (itch, pain, stinging, burning and skin tightness) and participant observable signs (skin dryness, cracking, scaling, shedding or flaking, redness and bleeding) using 0 to 10 numerical rating scales for severity. Two sub scores each ranging from 0 to 100 were derived: the psoriasis symptom score and the psoriasis sign score. A higher score indicated more severe disease.
Time Frame: Week 68
Population: For part 2, ITT analysis set included all randomized participants at Week 28 or treated with at least one dose of study agent within study part 2 (study group 2c) and those who had PSSD sign score >=1 at Week 28.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Part 2 Group 2a: Guselkumab 100 mg Q8W | Part 2 Group 2b: Guselkumab 100 mg Q16W | Part 2 Group 2c: Guselkumab 100 mg Q8W
Number analyzed (Participants) | 86 | 92 | 453
Percentage of participants | 30.2 [22.1 to 39.4] | 21.7 [14.9 to 30.0] | 14.8 [12.1 to 17.8]

14. Secondary Outcome: Groups 2a and 2b: Serum Trough Guselkumab Levels at Weeks 20, 28, 36 and 68
Description: Serum trough guselkumab levels at Weeks 20, 28, 36 were analyzed. Serum samples were analyzed to determine trough concentrations of guselkumab using a validated specific, and sensitive method. Week 28 data are presented in Part 2 arms (Groups 2a and 2b) as these groups were established at Week 28, however pre-Week 28 trough concentrations are also reported under these groups to assess potential differences between Part 1 PK characteristics.
Time Frame: At Weeks 20, 28, 36, 68
Population: For part 2, Pharmacokinetic (PK) Intent-to-treat analysis set included all randomized participants who had at least post baseline PK sample available. . Here, 'N' (number of participants analyzed) signifies number of participants evaluable for this outcome measure. Here 'n' (number analyzed) signifies number of participants analyzed at specified timepoints.
Measure: Mean (Standard Deviation); unit: micrograms/mL
Arm/Group | Part 2 Group 2a: Guselkumab 100 mg Q8W | Part 2 Group 2b: Guselkumab 100 mg Q16W
Number analyzed (Participants) | 147 | 145
micrograms/mL
  At Week 20 | 1.61 (0.989) | 1.60 (1.049)
  At Week 28: number analyzed (Participants) | 144 | 144
  At Week 28 | 1.58 (1.010) | 1.67 (1.076)
  At Week 36: number analyzed (Participants) | 143 | 139
  At Week 36 | 1.68 (1.062) | 0.38 (0.396)
  At Week 68: number analyzed (Participants) | 133 | 131
  At Week 68 | 1.56 (0.960) | 0.31 (0.377)

15. Secondary Outcome: Groups 2d and 3c: Percentage of Participants Who Were Re-Treated Due to Loss of Disease Control (PASI >5) and Regain Control of Disease (PASI <3) 24 Weeks After Start of Re-Treatment
Description: Percentage of participants who were re-treated due to loss of disease control (PASI >5) and regain control of disease (PASI <3) 24 weeks after start of re-treatment was reported. PASI was a system used for assessing and grading severity of psoriatic lesions and their response to therapy. In PASI, body was divided into 4 regions: head, trunk, upper extremities, and lower extremities. Each of these areas was assessed separately for percentage of area involved, which translates to numeric score that ranged from 0 (indicates no involvement) to 6 (90%-100% involvement), and for erythema, induration, and scaling, which were each rated on a scale of 0 to 4. PASI produced a numeric score that could range from 0 (no psoriasis) to 72 (maximum psoriasis). Higher score indicated more severe disease.
Time Frame: Week R0 up to Week R24
Population: Group 2d included the SRe participants who lost the disease control between Week 28 and 68, entered the re-treatment arm to receive guselkumab. Group 3c included SRe participants with fluctuating disease at Week 68 or loss of disease control at any other visit after Week 68, entered the re-treatment arm to receive guselkumab.
Measure: Number; unit: Percentage of participants
Groups:
- Part 2 Group 2d: Re-Treatment Guselkumab 100mg: Participants from Groups 2a and 2b who lost control of disease (PASI >=5) until Week 60 or were not eligible to enter withdrawal (PASI >=3) at Week 68 were re-treated as Group 2d, receiving guselkumab 100 mg at 0, 8, and 16weeks from entering Group 2d.
Arm/Group | Part 2 Group 2d: Re-Treatment Guselkumab 100mg | Part 3 Group 3c: Re-Treatment Guselkumab 100mg
Number analyzed (Participants) | 9 | 227
Percentage of participants | 88.8 [29.2 to 100.0] | 98.2 [95.5 to 99.5]

16. Secondary Outcome: Groups 1, 2a, 2b, 2c, 2d,3a, 3b, and 3c: Percentage of Participants With Adverse Events as a Measure of Safety and Tolerability
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of a medicinal (investigational or non-investigational) product, whether or not related to that medicinal (investigational or non-investigational) product.
Time Frame: Group 1: From Week 0 to Week 28; Group 2a,2b 2c: From Week 28 to Week 68; Group 3a, 3b: From Week 68 to Week 220; Group 2d, 3c: From Week R0 to Week R28
Population: ITT analysis set for part 1 included all participants treated with at least one dose of study agent. For part 2, ITT analysis set was used. For part 3, ITT analysis set included all participants entering study part 3. n=0, signifies that specified timepoint was not applicable for that arm. Here, 'N' (number of participants analyzed) signifies number of participants evaluable for this outcome measure. Here 'n' (number analyzed) signifies number of participants analyzed at specified timepoints.
Measure: Number; unit: Percentage of participants
Arm/Group | Part 1 Group 1: Guselkumab 100mg | Part 2 Group 2a: Guselkumab 100 mg Q8W | Part 2 Group 2b: Guselkumab 100 mg Q16W | Part 2 Group 2c: Guselkumab 100 mg Q8W | Part 2 Group 2d: Re-Treatment Guselkumab 100mg | Part 3 Group 3a: Withdrawal (Q8W) | Part 3 Group 3b: Withdrawal (Q16W) | Part 3 Group 3c: Re-Treatment Guselkumab 100mg
Number analyzed (Participants) | 880 | 148 | 149 | 525 | 9 | 136 | 137 | 236
Percentage of participants
  From Week 0 to Week 28: number analyzed (Participants) | 880 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  From Week 0 to Week 28 | 74.8 |  |  |  |  |  |  |
  From Week 28 to Week 68: number analyzed (Participants) | 0 | 148 | 149 | 525 | 0 | 0 | 0 | 0
  From Week 28 to Week 68 |  | 68.9 | 69.8 | 72.0 |  |  |  |
  Week 68 to Week 220: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 136 | 137 | 0
  Week 68 to Week 220 |  |  |  |  |  | 55.1 | 55.5 |
  From Week R0 to Week R28: number analyzed (Participants) | 0 | 0 | 0 | 0 | 9 | 0 | 0 | 236
  From Week R0 to Week R28 |  |  |  |  | 66.6 |  |  | 58.1

17. Secondary Outcome: Groups 1, 2a, 2b, 2c, 2d, 3a,3b and 3c: Number of Participants With Clinically Significant Laboratory Abnormalities
Description: Number of participants with clinically significant laboratory abnormalities was reported. Data of participants with at least one lab abnormality is reported. Abnormality criteria: Aspartate Aminotransferase (AST) >3, Alanine Aminotransferase (ALT).>5. For arm 3a and 3b, no drug was administered, hence no laboratory data was collected, per planned analysis.
Time Frame: Group 1: Week 20, Group 2a, 2b,2c: Week 68 and Group 2d and 3c: Week R28
Population: ITT analysis set for part 1 included all participants treated with at least one dose of study agent. For part 2, ITT analysis set included all randomized participants at week 28 or treated with at least one dose of study agent within study part 2 (study group 2c). For part 3, ITT analysis set included all participants entering study part 3. 'n' (number analyzed)=number of participants analyzed at specified timepoints. n=0 signifies that timepoint was not applicable for that arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 Group 1: Guselkumab 100mg | Part 2 Group 2a: Guselkumab 100 mg Q8W | Part 2 Group 2b: Guselkumab 100 mg Q16W | Part 2 Group 2c: Guselkumab 100 mg Q8W | Part 2 Group 2d: Re-Treatment Guselkumab 100mg | Part 3 Group 3c: Re-Treatment Guselkumab 100mg
Number analyzed (Participants) | 880 | 148 | 149 | 525 | 9 | 227
Participants
  AST > 3 (Week 20): number analyzed (Participants) | 880 | 0 | 0 | 0 | 0 | 0
  AST > 3 (Week 20) | 2 |  |  |  |  |
  ALT > 5 (Week 20): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
  AST > 3 (Week 68): number analyzed (Participants) | 0 | 148 | 149 | 525 | 9 | 0
  AST > 3 (Week 68) |  | 1 | 0 | 1 | 0 |
  ALT > 5 (Week 68): number analyzed (Participants) | 0 | 148 | 149 | 525 | 9 | 0
  ALT > 5 (Week 68) |  | 1 | 1 | 0 | 0 |
  AST > 3 (Week R28): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 227
  AST > 3 (Week R28) |  |  |  |  |  | 0
  ALT > 5 (Week R28): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 227
  ALT > 5 (Week R28) |  |  |  |  |  | 1

ADVERSE EVENTS:
Time Frame: Group 1: All-cause mortality: From screening (Week -4) to Week 28; serious and other AEs: Week0 to Week 28; Groups 2a,2b,2c (all-cause mortality and SAEs/other AEs): Week 28 to Week 68; Groups 3a, 3b (all-cause mortality and SAEs/other AEs): Week 68 to Week 220; Groups 2d, 3c (all-cause mortality and SAEs/other AEs): Week R0 to Week R28
Description: Same event may appear as AE and serious adverse event (SAE), what is presented are distinct events. Event may be categorized as serious in 1 participant and as non-serious in another subject or 1 participants may have experienced both serious and non-serious event during study. Safety analysis population included all participants who were treated with at least one dose of study drug. All-cause mortality population included all randomized subject.
Groups:
- Group 2a: Guselkumab 100 mg Q8W: Super responders (SRe) (Psoriasis Area and Severity Index [PASI] score = 0 at Week 20 and Week 28) who completed study Part 1, were randomized to receive guselkumab 100 mg by SC injection every 8 weeks (Q8W) starting at Week 28 until Week 60. Participants were followed from Week 28 until Week 68 or early termination prior to Week 68.
- Group 2b: Guselkumab 100 mg Q16W: Super responders (PASI score = 0 at Week 20 and Week 28) who completed study Part 1, were randomized to receive guselkumab 100 mg by SC injection every 16 weeks (Q16W) at Weeks 36 and 52. To maintain the study blind, participants were administered placebo by SC injection at Weeks 28, 44 and 60. Participants were followed from Week 28 until Week 68 or early termination prior to Week 68.
- Group 2c: Guselkumab 100 mg Q8W: Non-super responders (PASI score greater than [>] 0 at Week 20 and/or Week 28) who completed study Part 1 continued to receive guselkumab 100 mg by SC injection Q8W starting at Week 28 till Week 60. Participants were followed from Week 28 until Week 68 or early termination prior to Week 68.
- Group 3a Guselkumab 100 mg Q8W: Super responders from Group 2a with PASI score <= 3 were withdrawn from guselkumab 100 mg by SC injection every 8 weeks (Q8W) at Week 68. Participants were followed until Week 220.
- Group 3b Guselkumab 100 mg Q16W: Super responders from Group 2b with PASI score <= 3 who were withdrawn from guselkumab 100 mg by SC injection every 16 weeks (Q16W) at Week 68. Participants were followed until Week 220.
- Group 3c Guselkumab 100 mg: Super responders with loss of disease control at or any visit after week 68 who entered the re-treatment arm and received guselkumab 100 mg by SC injection at re-treatment weeks 0, 8 and 16 calculated from the date of loss of disease control. Participants were followed from Week 0 until Week 24 calculated from start of re-treatment due to loss disease control.
Arm/Group | Part 1 Group 1: Guselkumab 100mg | Group 2a: Guselkumab 100 mg Q8W | Group 2b: Guselkumab 100 mg Q16W | Group 2c: Guselkumab 100 mg Q8W | Part 2 Group 2d: Re-Treatment Guselkumab 100mg | Group 3a Guselkumab 100 mg Q8W | Group 3b Guselkumab 100 mg Q16W | Group 3c Guselkumab 100 mg
All-Cause Mortality (participants affected / at risk) | 1/880 | 0/148 | 0/150 | 1/525 | 0/9 | 0/136 | 0/137 | 0/227
Serious Adverse Events (participants affected / at risk) | 38/880 | 7/148 | 6/149 | 33/525 | 0/9 | 3/136 | 9/137 | 8/227
Other Adverse Events (participants affected / at risk) | 631/880 | 101/148 | 103/149 | 367/525 | 6/9 | 75/136 | 75/137 | 130/227
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 Group 1: Guselkumab 100mg (N=880) | Group 2a: Guselkumab 100 mg Q8W (N=148) | Group 2b: Guselkumab 100 mg Q16W (N=149) | Group 2c: Guselkumab 100 mg Q8W (N=525) | Part 2 Group 2d: Re-Treatment Guselkumab 100mg (N=9) | Group 3a Guselkumab 100 mg Q8W (N=136) | Group 3b Guselkumab 100 mg Q16W (N=137) | Group 3c Guselkumab 100 mg (N=227)
Splenic Haematoma (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute Coronary Syndrome (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute Myocardial Infarction (Cardiac disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Arteriosclerosis Coronary Artery (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cardiac Failure Chronic (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Coronary Artery Disease (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1
Myocarditis (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal Hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colitis Ischaemic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hiatus Hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chest Pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis Chronic (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anaphylactic Reaction (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Autoimmune Disorder (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abscess of External Auditory Meatus (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anal Abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Bacterial Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chronic Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Covid-19 (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infectious Mononucleosis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Peritonsillar Abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post Procedural Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcal Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tooth Abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ankle Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Bone Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cartilage Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Clavicle Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Foot Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Humerus Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ligament Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ligament Rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pelvic Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Radius Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rib Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seroma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Traumatic Liver Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Benign Hepatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Colorectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Craniopharyngioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Squamous Cell Carcinoma of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tumour Haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cerebellar Infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cerebral Infarction (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebrovascular Accident (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nerve Compression (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Polyneuropathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pseudoradicular Syndrome (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Transient Ischaemic Attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Mental Disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Suicidal Behaviour (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ovarian Cyst (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypersensitivity Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aortic Aneurysm (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Extremity Necrosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertensive Urgency (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 Group 1: Guselkumab 100mg (N=880) | Group 2a: Guselkumab 100 mg Q8W (N=148) | Group 2b: Guselkumab 100 mg Q16W (N=149) | Group 2c: Guselkumab 100 mg Q8W (N=525) | Part 2 Group 2d: Re-Treatment Guselkumab 100mg (N=9) | Group 3a Guselkumab 100 mg Q8W (N=136) | Group 3b Guselkumab 100 mg Q16W (N=137) | Group 3c Guselkumab 100 mg (N=227)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 4 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Splenomegaly (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Spontaneous Haematoma (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Angina Pectoris (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Aortic Valve Incompetence (Cardiac disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Aortic Valve Sclerosis (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Aortic Valve Stenosis (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cardiac Failure (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cardiac Perfusion Defect (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cardiovascular Disorder (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Coronary Artery Disease (Cardiac disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Heart Valve Incompetence (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Left Ventricular Hypertrophy (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Mitral Valve Incompetence (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sinus Tachycardia (Cardiac disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Supraventricular Extrasystoles (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 4 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Epidermal Naevus (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gilbert's Syndrome (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Keratosis Follicular (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Phimosis (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Conductive Deafness (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deafness (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ear Pain (Ear and labyrinth disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ear Pruritus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Excessive Cerumen Production (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sudden Hearing Loss (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Androgen Deficiency (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Goitre (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hyperprolactinaemia (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Blepharitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Borderline Glaucoma (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chalazion (Eye disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Conjunctival Irritation (Eye disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Conjunctivitis Allergic (Eye disorders) | 4 | 1 | 0 | 0 | 0 | 2 | 0 | 0
Dry Eye (Eye disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eczema Eyelids (Eye disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Eye Irritation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eye Pruritus (Eye disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Eyelid Disorder (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Glaucoma (Eye disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Keratitis (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lacrimation Increased (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ocular Discomfort (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ocular Hyperaemia (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ocular Hypertension (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Optic Nerve Disorder (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Retinal Haemorrhage (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ulcerative Keratitis (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vision Blurred (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Visual Acuity Reduced (Eye disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Visual Impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 3 | 3 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal Distension (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal Hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 6 | 0 | 1 | 4 | 0 | 0 | 0 | 0
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 4 | 1 | 0 | 9 | 0 | 0 | 0 | 2
Anal Fissure (Gastrointestinal disorders) | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Aphthous Ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Colitis Ischaemic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dental Caries (Gastrointestinal disorders) | 3 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Dental Discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dental Necrosis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 24 | 5 | 1 | 13 | 0 | 1 | 0 | 5
Diverticulum Intestinal (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dry Mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 3 | 0 | 1 | 3 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Epigastric Discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erosive Duodenitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Faeces Soft (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 2 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Food Poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastric Disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 4 | 0 | 0 | 2 | 0 | 0 | 0 | 1
Gastrointestinal Disorder (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal Pain (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastrointestinal Polyp Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 4 | 0 | 0 | 1 | 0 | 1 | 1 | 1
Gingival Bleeding (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gingival Cyst (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gingival Recession (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoids Thrombosed (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hiatus Hernia (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Inguinal Hernia (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Large Intestine Polyp (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mouth Cyst (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 14 | 2 | 1 | 4 | 0 | 1 | 0 | 2
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Paraesthesia Oral (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Periodontal Disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Poor Dental Condition (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rectal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tongue Discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 5 | 0 | 1 | 3 | 0 | 0 | 1 | 2
Umbilical Hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 8 | 0 | 1 | 3 | 0 | 0 | 0 | 2
Adverse Drug Reaction (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Application Site Erythema (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chest Discomfort (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chest Pain (General disorders) | 6 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cyst (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug Ineffective (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 14 | 1 | 2 | 4 | 0 | 1 | 0 | 0
Foreign Body Reaction (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
General Physical Health Deterioration (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Impaired Healing (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza Like Illness (General disorders) | 3 | 1 | 1 | 0 | 0 | 0 | 1 | 2
Injection Site Erythema (General disorders) | 8 | 6 | 0 | 5 | 0 | 0 | 0 | 2
Injection Site Haematoma (General disorders) | 2 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Injection Site Hypersensitivity (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injection Site Induration (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injection Site Oedema (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Injection Site Pain (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Injection Site Paraesthesia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Injection Site Pruritus (General disorders) | 2 | 2 | 0 | 4 | 0 | 0 | 0 | 0
Injection Site Reaction (General disorders) | 2 | 1 | 0 | 5 | 0 | 0 | 0 | 0
Injection Site Scar (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection Site Swelling (General disorders) | 3 | 1 | 0 | 1 | 0 | 0 | 0 | 2
Localised Oedema (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oedema Peripheral (General disorders) | 6 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pain (General disorders) | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Peripheral Swelling (General disorders) | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 4 | 3 | 1 | 3 | 0 | 1 | 1 | 1
Temperature Intolerance (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaccination Site Erythema (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaccination Site Pain (General disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0
Biliary Colic (Hepatobiliary disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Hepatic Steatosis (Hepatobiliary disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Hepatosplenomegaly (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Allergy to Arthropod Bite (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Allergy to Arthropod Sting (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anaphylactic Reaction (Immune system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Contrast Media Reaction (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Food Allergy (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Mite Allergy (Immune system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Seasonal Allergy (Immune system disorders) | 4 | 0 | 1 | 1 | 0 | 0 | 1 | 1
Abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abscess Jaw (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abscess Limb (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abscess Oral (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acarodermatitis (Infections and infestations) | 3 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Acne Pustular (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute Sinusitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anal Abscess (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Bacterial Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bacterial Vaginosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Balanitis Candida (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Body Tinea (Infections and infestations) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Borrelia Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Breast Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 12 | 1 | 1 | 10 | 0 | 3 | 2 | 2
Bronchitis Bacterial (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Candida Infection (Infections and infestations) | 1 | 0 | 0 | 4 | 0 | 0 | 0 | 0
Cervicitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chronic Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 4 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Coronavirus Infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 2 | 3 | 2
Covid-19 (Infections and infestations) | 10 | 4 | 3 | 13 | 1 | 20 | 12 | 21
Cystitis (Infections and infestations) | 9 | 1 | 1 | 2 | 0 | 0 | 0 | 0
Dermatitis Infected (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dermatophytosis of Nail (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diabetic Foot Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Ear Infection (Infections and infestations) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eczema Infected (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enteritis Infectious (Infections and infestations) | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Epididymitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 3 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Erythema Migrans (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 7 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Fungal Foot Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Fungal Infection (Infections and infestations) | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Fungal Skin Infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0
Furuncle (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastric Ulcer Helicobacter (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 18 | 1 | 1 | 3 | 0 | 0 | 2 | 3
Gastroenteritis Clostridial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastroenteritis Viral (Infections and infestations) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal Infection (Infections and infestations) | 12 | 1 | 2 | 9 | 0 | 0 | 1 | 0
Gastrointestinal Viral Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Genital Candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Genital Herpes (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Genital Infection Bacterial (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Genital Infection Fungal (Infections and infestations) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Gingivitis (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Hantaviral Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Helicobacter Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes Simplex (Infections and infestations) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Herpes Virus Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes Zoster (Infections and infestations) | 6 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 4 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Infected Bite (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infected Cyst (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infected Dermal Cyst (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infected Skin Ulcer (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infectious Mononucleosis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infective Glossitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 8 | 5 | 5 | 6 | 0 | 1 | 2 | 1
Joint Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Localised Infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lyme Disease (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Malassezia Infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Mastitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nail Bed Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasal Herpes (Infections and infestations) | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 214 | 26 | 23 | 97 | 0 | 17 | 17 | 32
Oesophageal Candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Onychomycosis (Infections and infestations) | 5 | 1 | 0 | 3 | 0 | 1 | 1 | 2
Oral Candidiasis (Infections and infestations) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Oral Fungal Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Oral Herpes (Infections and infestations) | 8 | 2 | 3 | 6 | 0 | 0 | 2 | 0
Otitis Externa (Infections and infestations) | 4 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Otitis Media (Infections and infestations) | 1 | 1 | 0 | 3 | 1 | 0 | 0 | 0
Otitis Media Viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paronychia (Infections and infestations) | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0
Parotitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic Inflammatory Disease (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Periodontitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Peritonsillar Abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Post Procedural Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Post-Acute Covid-19 Syndrome (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Postoperative Wound Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulpitis Dental (Infections and infestations) | 4 | 1 | 2 | 4 | 0 | 1 | 0 | 2
Pustule (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pyelitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Respiratory Tract Infection (Infections and infestations) | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 13 | 0 | 1 | 4 | 0 | 0 | 2 | 2
Root Canal Infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Scarlet Fever (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 8 | 3 | 1 | 4 | 0 | 1 | 5 | 2
Skin Bacterial Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin Candida (Infections and infestations) | 4 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Skin Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcal Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Subcutaneous Abscess (Infections and infestations) | 1 | 0 | 2 | 1 | 0 | 1 | 0 | 0
Tinea Cruris (Infections and infestations) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Tinea Infection (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Tinea Manuum (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tinea Pedis (Infections and infestations) | 5 | 4 | 1 | 6 | 0 | 0 | 1 | 1
Tinea Versicolour (Infections and infestations) | 2 | 1 | 0 | 2 | 0 | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 12 | 2 | 3 | 6 | 0 | 0 | 1 | 3
Tonsillitis Bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth Abscess (Infections and infestations) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Tooth Infection (Infections and infestations) | 4 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 22 | 1 | 0 | 3 | 0 | 1 | 1 | 4
Urethritis Gonococcal (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 8 | 1 | 3 | 4 | 1 | 1 | 1 | 1
Urinary Tract Infection Bacterial (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Vaginal Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Viral Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Viral Rash (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Viral Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal Mycotic Infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Wound Infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ankle Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Arthropod Bite (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Arthropod Sting (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Bone Contusion (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 2 | 0 | 0 | 2 | 2
Burns Second Degree (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Burns Third Degree (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chemical Burn of Skin (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chillblains (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Clavicle Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 6 | 4 | 4 | 4 | 0 | 0 | 0 | 1
Corneal Abrasion (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Epicondylitis (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Eye Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eye Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fibula Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Foot Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Foreign Body in Eye (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fractured Coccyx (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hand Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0
Heat Stroke (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Human Bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Humerus Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Inappropriate Schedule of Product Administration (Injury, poisoning and procedural complications) | 11 | 2 | 4 | 14 | 0 | 0 | 0 | 3
Incision Site Erythema (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Incomplete Spinal Fusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint Capsule Rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Joint Dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Joint Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ligament Rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 2 | 0 | 0 | 2 | 2
Ligament Sprain (Injury, poisoning and procedural complications) | 4 | 1 | 3 | 4 | 0 | 1 | 1 | 0
Limb Injury (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 4 | 0 | 0 | 1 | 2
Lower Limb Fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Meniscus Injury (Injury, poisoning and procedural complications) | 3 | 1 | 0 | 5 | 0 | 0 | 0 | 0
Muscle Rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Muscle Strain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post Procedural Hypothyroidism (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Post Procedural Swelling (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Post-Traumatic Pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Procedural Dizziness (Injury, poisoning and procedural complications) | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Procedural Pain (Injury, poisoning and procedural complications) | 6 | 1 | 1 | 4 | 0 | 1 | 0 | 1
Rib Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Road Traffic Accident (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin Abrasion (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin Laceration (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tendon Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tendon Rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Thermal Burn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tooth Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Traumatic Haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary Retention Postoperative (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vaccination Complication (Injury, poisoning and procedural complications) | 2 | 1 | 4 | 6 | 0 | 4 | 0 | 5
Wound (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 3 | 0 | 1 | 0 | 0
Wrist Fracture (Injury, poisoning and procedural complications) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 7 | 3 | 2 | 3 | 0 | 0 | 0 | 2
Aortic Bruit (Investigations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Aspartate Aminotransferase Abnormal (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate Aminotransferase Increased (Investigations) | 2 | 1 | 0 | 2 | 0 | 0 | 0 | 2
Basophil Count Increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bilirubin Conjugated Increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood Bilirubin Increased (Investigations) | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 1
Blood Bilirubin Unconjugated Increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood Cholesterol Increased (Investigations) | 4 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Blood Creatine Phosphokinase Abnormal (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood Creatine Phosphokinase Increased (Investigations) | 20 | 3 | 6 | 8 | 0 | 1 | 0 | 7
Blood Creatinine Increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood Glucose Decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood Glucose Increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood Lactate Dehydrogenase Increased (Investigations) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood Potassium Abnormal (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood Potassium Increased (Investigations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood Pressure Increased (Investigations) | 2 | 1 | 0 | 1 | 0 | 0 | 2 | 0
Blood Triglycerides Increased (Investigations) | 11 | 0 | 0 | 4 | 0 | 0 | 0 | 4
Blood Urea Increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood Uric Acid Increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Body Temperature Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cardiac Murmur (Investigations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gamma-Glutamyltransferase Increased (Investigations) | 9 | 3 | 1 | 4 | 0 | 0 | 0 | 1
Glycosylated Haemoglobin Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haematocrit Increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Heart Rate Increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Hepatic Enzyme Increased (Investigations) | 4 | 1 | 1 | 3 | 0 | 0 | 0 | 3
Lipase Increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lipids Increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Liver Function Test Increased (Investigations) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 1
Lymphocyte Count Decreased (Investigations) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Lymphocyte Morphology Abnormal (Investigations) | 3 | 0 | 0 | 3 | 0 | 0 | 0 | 2
Neutrophil Count Decreased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neutrophil Count Increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Platelet Count Decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Platelet Count Increased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Prostatic Specific Antigen Increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spermatozoa Abnormal (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Streptococcus Test Positive (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Transaminases Increased (Investigations) | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 1
Tri-Iodothyronine Free Increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight Decreased (Investigations) | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Weight Increased (Investigations) | 4 | 0 | 0 | 1 | 0 | 0 | 0 | 0
White Blood Cell Count Increased (Investigations) | 2 | 0 | 0 | 3 | 0 | 0 | 0 | 0
White Blood Cell Morphology Abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diabetes Mellitus (Metabolism and nutrition disorders) | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fat Intolerance (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 5 | 1 | 0 | 3 | 0 | 1 | 1 | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 3 | 0 | 0 | 0 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 4 | 0 | 0 | 2 | 0 | 0 | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 5 | 1 | 0 | 2 | 0 | 0 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypovitaminosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Selenium Deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 3 | 1 | 0 | 3 | 0 | 0 | 0 | 0
Vitamin B12 Deficiency (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Vitamin D Deficiency (Metabolism and nutrition disorders) | 1 | 2 | 0 | 2 | 0 | 1 | 2 | 0
Weight Fluctuation (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 41 | 4 | 5 | 29 | 0 | 8 | 4 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 26 | 6 | 8 | 13 | 1 | 4 | 2 | 3
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 0 | 1 | 1 | 0
Chondropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dactylitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Enthesopathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Extremity Contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Groin Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Intervertebral Disc Degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 2 | 3 | 0 | 6 | 0 | 0 | 2 | 0
Jaw Disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Joint Stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint Swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Limb Discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscle Tightness (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal Discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 2 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 2 | 0 | 3 | 0 | 0 | 0 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Nodal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Osteitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 9 | 0 | 0 | 3 | 0 | 1 | 1 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 6 | 0 | 3 | 6 | 0 | 0 | 1 | 5
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Plantar Fasciitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Polymyalgia Rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Psoriatic Arthropathy (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0 | 6 | 0 | 0 | 1 | 0
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 0
Sacral Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tendon Disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Trigger Finger (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anogenital Warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 2 | 0 | 1 | 0 | 1
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Benign Hepatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Benign Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Benign Neoplasm of Adrenal Gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Benign Neoplasm of Eyelid (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysplastic Naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Fibroadenoma of Breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Fibrous Histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Melanocytic Naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 2 | 1 | 3 | 0 | 1 | 0 | 0
Osteoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seborrhoeic Keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 3 | 2 | 0 | 0 | 1 | 0
Squamous Cell Carcinoma of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ageusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anosmia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Carpal Tunnel Syndrome (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebellar Stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cervicobrachial Syndrome (Nervous system disorders) | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cognitive Disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cubital Tunnel Syndrome (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Disturbance in Attention (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 1 | 2 | 0 | 1 | 0 | 2
Dizziness Postural (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Facial Paralysis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gliosis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Head Discomfort (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 79 | 8 | 9 | 29 | 0 | 6 | 3 | 13
Hypoaesthesia (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Loss of Consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Migraine (Nervous system disorders) | 6 | 2 | 2 | 1 | 0 | 0 | 1 | 0
Migraine with Aura (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nerve Compression (Nervous system disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neuritis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neuropathy Vitamin B6 Deficiency (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Orthostatic Intolerance (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Peripheral Nerve Lesion (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post Herpetic Neuralgia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Precerebral Arteriosclerosis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pseudoradicular Syndrome (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Radiculopathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Restless Legs Syndrome (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 3 | 1 | 1 | 3 | 0 | 0 | 0 | 0
Sensory Disturbance (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 1
Tension Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Thoracic Outlet Syndrome (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thoracic Radiculopathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 2 | 1 | 2 | 2 | 0 | 0 | 0 | 1
Device Physical Property Issue (Product Issues) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Attention Deficit Hyperactivity Disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Burnout Syndrome (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 4 | 0 | 0 | 1 | 0 | 1 | 2 | 2
Depressive Symptom (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 0 | 0 | 2 | 0 | 1 | 0 | 0
Panic Attack (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Personality Disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Post-Traumatic Stress Disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Restlessness (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sleep Disorder (Psychiatric disorders) | 3 | 0 | 0 | 2 | 0 | 0 | 1 | 1
Sleep Disorder Due to A General Medical Condition (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stress (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Suicidal Behaviour (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nephritis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urethral Stenosis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary Incontinence (Renal and urinary disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 3 | 0 | 0 | 2 | 0 | 0 | 1 | 0
Endometriosis (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erectile Dysfunction (Reproductive system and breast disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhagic Ovarian Cyst (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Heavy Menstrual Bleeding (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Menopausal Symptoms (Reproductive system and breast disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Menstruation Irregular (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ovarian Cyst (Reproductive system and breast disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Polycystic Ovaries (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Prostatomegaly (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus Genital (Reproductive system and breast disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Testicular Torsion (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal Dryness (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Allergic Respiratory Symptom (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Allergic Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 2 | 0 | 0 | 0 | 0
Catarrh (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 4 | 2 | 10 | 0 | 4 | 1 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypersensitivity Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Increased Upper Airway Secretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Larynx Irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal Discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasal Pruritus (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Nasal Septum Deviation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 12 | 1 | 0 | 5 | 0 | 1 | 1 | 2
Painful Respiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 1 | 0 | 1 | 0 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Tonsillar Disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper Airway Obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 3 | 1 | 1 | 3 | 0 | 1 | 0 | 0
Actinic Keratosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 5 | 1 | 0 | 3 | 0 | 0 | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chloasma (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermal Cyst (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 5 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Dermatitis Psoriasiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug Eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 0 | 0 | 1 | 1 | 0
Dyshidrotic Eczema (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 8 | 1 | 0 | 11 | 0 | 0 | 0 | 1
Eczema Asteatotic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eczema Nummular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Erythema Nodosum (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythrodermic Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 5 | 1 | 1 | 3 | 0 | 0 | 0 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ingrowing Nail (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Intertrigo (Skin and subcutaneous tissue disorders) | 11 | 0 | 0 | 1 | 0 | 1 | 1 | 1
Koebner Phenomenon (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nail Dystrophy (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nail Psoriasis (Skin and subcutaneous tissue disorders) | 4 | 0 | 3 | 5 | 0 | 3 | 0 | 4
Night Sweats (Skin and subcutaneous tissue disorders) | 5 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Perioral Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Photosensitivity Reaction (Skin and subcutaneous tissue disorders) | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pityriasis Rosea (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Polymorphic Light Eruption (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Prurigo (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 9 | 2 | 3 | 5 | 0 | 5 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 17 | 1 | 1 | 8 | 0 | 10 | 12 | 7
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Rash Erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash Pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Seborrhoeic Dermatitis (Skin and subcutaneous tissue disorders) | 6 | 1 | 1 | 1 | 0 | 0 | 1 | 0
Skin Burning Sensation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin Disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin Fissures (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin Fragility (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin Induration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin Irritation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin Maceration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin Mass (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin Texture Abnormal (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Solar Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Stasis Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Toxic Skin Eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 5 | 1 | 0 | 7 | 0 | 1 | 0 | 0
Urticaria Contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urticaria Physical (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Vitiligo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Stress at Work (Social circumstances) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood Pressure Fluctuation (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Extremity Necrosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Hot Flush (Vascular disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 48 | 4 | 5 | 31 | 0 | 3 | 3 | 7
Hypertensive Crisis (Vascular disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Hypertensive Urgency (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Peripheral Arterial Occlusive Disease (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Peripheral Venous Disease (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Thrombophlebitis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Varicose Vein (Vascular disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
White Coat Hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nail psoriasis (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pruritus genital (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
There was an interruption of enrollment due to Corona Pandemic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2024-09-26): https://cdn.clinicaltrials.gov/large-docs/35/NCT03818035/Prot_002.pdf
  • Statistical Analysis Plan (2025-04-23): https://cdn.clinicaltrials.gov/large-docs/35/NCT03818035/SAP_003.pdf